CLINICAL TRIAL: NCT05222282
Title: Sexual Health in Patients With Hematologic Malignancies - Symptom Assessment and Management
Brief Title: Sexual Health in Patients With Hematologic Malignancies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Kristina Holmegaard Nørskov, Clinical Nurse Specialist, PhD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Sexual Health
Record Dates: First submitted 2021-12-15; First posted 2022-02-03 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Sexuality; Sexual Dysfunction; Psychological; Quality of Life; Symptoms and Signs
Keywords: sexual health; hematologic malignancy; sexual dysfunction; quality of life; symptom assessment; symptom management
MeSH Terms: conditions — Sexuality; Sexual Dysfunction, Physiological; Signs and Symptoms; Hematologic Neoplasms | interventions — Sexual Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention with
  1. nurseled sexual consultations with screening questionnaire prior to consultation
  2. genital examintaion with doctor
  Interventions: Other: Sexual Health
- Kontrol (Other): Usual care
  Interventions: Other: Sexual Health

INTERVENTIONS:
Other: Sexual Health — Prevention of sexual dysfunction

SUMMARY:
Sexual wellbeing is an integral component of psychosocial and physical wellbeing. Cancer-related symptoms, treatment side-effects and psychosocial distress have significant impact on sexual well-being and sexual health. Within the framework of sexual wellbeing, sexual function is defined by a capacity to fully engage in all phases of the human sexual response cycle. Thus, sexual dysfunction is characterized by a disruption in one or more elements of the response cycle. Previous research shows that patients with hematologic malignancies and specifically patients following stem cell transplantation experience a high symptom burden and distinct genital alterations, and therefore in increased risk of sexual dysfunction. In spite of growing evidence documenting high prevalence of sexual dysfunction in cancer patients, patients with hematologic malignancies are underrepresented in clinical trials investigating their sexual health. This study aims to examine the sexual health in patients across hematologic malignancies in Denmark, and to investigate feasiblity and effect of a randomized multimodal intervention by providing nurse-led sexual consultations and physician-led preventive genital examinations, to enhance sexual function and early recognition of gential graft versus host disease in adult patients following hematopoietic stem cell transplantation. Finally, the study aims to explore perspectives and experiences of patients following this multimodal intervention. This knowledge will entail new opportunities to detect subgroups of patients with distinct risk of sexual dysfunction, and potentially lead to targeted interventions in clinical practice toward this specific population. Moreover this will provide evidence with high methodological rigor and potentially strengthen the possibilities for evidence-based decision making in Denmark regarding preventive gential examinations during follow-up in patients following stem cell transplant.

DETAILED DESCRIPTION:
1. Introduction As the survival rates for hematologic malignancies improves there is subsequently an increased need for addressing long-term complications. The evidence highlight that patients experience a high symptom burden including sexual dysfunction, and therefore in increased risk of decreased sexual health. Sexual health is a state of physical, mental and social well-being in relation to sexuality, and can reduce the emotional distress and improve psychosocial response to a cancer diagnosis and complications following treatment. Still, this population is underrepresented in clinical trials investigating their sexual health. It is therefore essential to include them in future clinical trials in order to have a comprehensive view of their condition of sexual health and sexual function. This knowledge will entail new opportunities to detect subgroups of patients with distinct risk of sexual dysfunction, and this will potentially lead to targeted interventions in clinical practice toward this specific population.

   In patients with hematologic malignancies undergoing hematopoietic stem cell transplantation (HSCT) sexual dysfunction is one of the most frequent long-term issues. Sexual dysfunction include decreased libido, vaginal alterations, erectile and ejaculatory dysfunction, dysfunction in sexual hormones, dyspareunia and infertility. Specifically, an immunologic reaction in the skin tissue called genital graft versus host disease (GHVD), is a major determinant of sexual dysfunction in this population. Genital GVHD can lead to vaginal stenosis, scar tissue and adhesions in blood vessels, rash and increased sensitivity in the skin of the genitals. Despite increasing evidence on the clinical manifestations it is still an underrecognized and underestimated complication of HCST in clinical practice due to the nonspecific nature of presenting symptoms and low awareness of the condition. In a previous systematic review, the investigators concluded that multiple aspects of sexuality were affected following treatment with HSCT, and the impact and ethology of these sexual alterations were different between genders. Therefore, the investigators investigated the impact of HSCT on sexuality in a resent longitudinal survey. The results showed a significant decline in overall sexual function in both men and women. Still, most studies have solely investigated female genital GVHD, in small populations and only few have included evaluations of sexual function prior to HSCT. No previous studies have investigated the effect of a multimodal intervention specifically focused on evaluation of sexual function through nurse-led sexual consultations and early recognition of genital GVHD in patients during treatment with HSCT. Thus, further recognition of sexual symptoms and regular follow-up can possibly help to improve the detection and facilitate early treatment of sexual complications including genital GVHD. This will help our understanding in the development of systematic strategies to prevent or treat its long-term effects.
2. Hypotheses

   This study is based on the following hypothesis or assumptions:

   Study 1

   • The investigators hypothesize that patients with hematologic malignancies report impaired sexual function, and that sexual dysfunction are associated with high symptom burden, sexual distress, reduced quality of life and increased anxiety and depression.

   Study 2

   • The investigators hypothesize that a multimodal intervention with nurse-led sexual counseling and systematic gential evaluations is feasible and will enhance sexual function in patients undergoing HSCT
3. Aim The overall aim of this study is to investigate sexual health in patients treated for a hematologic malignancy, and to generate research-based knowledge on the feasiblity and effect of a multimodal intervention with nurse-led sexual counseling and systematic genital evaluation on sexual function in patients during their treatment with HSCT.

   The specific aims of the studies are:

   Study 1

   • To examine the sexual health in patients across hematologic malignancies in Denmark, and to examine the prevalence and factors associated with sexual dysfunction in this population.

   Study 2

   • To investigate feasibility and effect of a randomized multimodal intervention with nurse-led sexual counseling and systematic genital evaluation on enhancing sexual function in patients undergoing HSCT.
4. Study description study 1 4.1 Aim To examine the sexual health in patients across hematologic malignancies in Denmark, and to examine the prevalence and factors associated with sexual dysfunction in this population.

   4.2 Design and methods This study is an explorative cross-sectional national study examining sexual health across different haematological malignant diseases in Denmark.

   4.3 Participants Participants with haematological malignant diseases specifically acute myeloid leukemia (AML), acute lymphatic leukemia (ALL), chronic lymphatic leukemia (CLL), chronic myeloid leukemia (CML), multiple myeloma, non-Hodgkin lymphoma, Hodgkin lymphoma, are eligible if > 18 years with time post diagnosis > 3 month up to 10 years. Participants are excluded if they are unable to read or speak Danish or have a cognitive disorder.

   4.4 Recruitment and procedure Eligible participants will be identified through the National Patient Register. Then, the Danish Health Data Authority will be applied to extract a representative sample from the full potential eligible participants. This sample will be based on statistical measurements to achieve high statistical power. Eligible participants will receive information about the study, provide written informed consent and receive the questionnaires electronically through e-boks.

   4.5 Data collection

   Participant and disease characteristics will be obtained from the participants. These will include age, gender, marital status, education, employment status, disease type and status, type and intensity of treatment received, and treated hospital. The patient-reported outcome measure (PROM) include:
   * Sexual health will be assessed by the Female Sexual Function Index (FSFI) in female participants. FSFI is a brief 19-item self-report measure of female sexual function that provides scores on six domains: desire, arousal, lubrication, orgasm, satisfaction and pai. In male participants, sexual health will be assessed by The International Index of Erectile Function Questionnaire (IIEF). IIEF is a brief 15-item widely used multi-dimensional self-report instrument for evaluation of male sexual function that proves scores in five domains: erectile function, orgasmic function, sexual desire, intercourse satisfaction, and overall satisfaction.
   * Sexual distress will be assessed by the Female Sexual Distress Scale - Revised (FSDS-R). FSDS-R is a 13 item measure assess sexual distress specifically related to low sexual desire. The scale has been developed for use in female patients but have recently been validated in male patients with excellent internal consistency and test-retest reliabilities.
   * Quality of life will be assessed by The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-C30). EORTC-C30 is a 30 item multi-dimensional quality of life measure designed for use in cancer patients.
   * Symptom burden will be assessed with M.D. Anderson Symptom Inventory (MDASI) which is a 19 item measure and assesses the severity of 13 symptoms and their impact in cancer patients.
   * Psychological well-being will be assessed and measured by using the Hospital Anxiety and Depression Scale (HADS), which is a brief 14-item self-report measure of anxiety and depression.

   4.6 Analysis Statistical analysis will be conducted using IBM SPSS Statistics for Windows, version 25. Throughout, two-sided P-values <0.05 confidence intervals are considered indicators of statistical significance.
5. Study description study 2 5.1. Aim To investigate feasibility and effect of a randomized multimodal intervention with nurse-led sexual counseling and systematic gential evaluation on enhancing sexual function in patients undergoing HSCT.

   5.2 Design and methods This study is a prospective two-arms randomized controlled trial to assess the feasibility and effect of a multimodal nonpharmacological intervention to address sexual health in patients undergoing HSCT.

   5.3 Participants Patients (age>18 years) with a hematologic malignancy who is planned to undergo an HSCT, who provide informed written consent and can understand, speak and read Danish are eligible to participate. The exclusion criteria include patients with dementia, psychotic disorders, or other cognitive diseases or conditions that hinder participation.

   5.4 Recruitment and procedure Patients will be recruited from the Department of Hematology, Rigshospitalet. Eligible participants receive oral and written project information from primary research investigator (KHN) during their preexamination week prior to HSCT. Patients will be informed about the trial, perceived benefits, risks, and safety precautions, and about their personal rights in entering the trial. Study participants who complete baseline questionnaires are then randomized, and participants in the intervention group will be scheduled for their first assessment.

   Randomization and blinding Patients included in the study will be randomized 1:1 ratio to either the intervention group or control group (usual care) by KHN. Randomization and stratification (age, diagnosis) will be performed through the randomization module in Redcap. Because it is not feasible, the primary investigator and the patient will not be blinded to group allocation. However, to reduce the risk of detection bias, the investigator will be blinded to group allocation during data entry. Moreover, the statistician will be blinded to allocation during data analysis. The identity of each patient will be masked and can only be re-identified using a separately kept key file.

   Usual care Patients allocated to control group will receive usual care which include genital evaluation during their preexamination week prior to HSCT. During the treatment trajectory genital examination is conducted when genital symptoms are reported either by the health care provider or the patient. Patients in the control arm will receive a final assessment with genital evaluation and nurse-led sexual counseling. Data collection with PROM will be conducted prior to the final genital evaluation and nurse-led sexual counseling.

   5.5 Multimodal Sexual Dysfunction Intervention The intervention consists of nurse-led sexual counselling and systematic genital evaluation (Figure 1). The intervention begins during their preexamination week prior to HSCT and the subsequent 18 months.

   Nurse-led sexual counseling The intervention entails five nurse-led sexual counseling sections. Participants will attend their first nurse-led sexual counseling session three month post HSCT with KHN who is an experienced HSCT nurse. The patients will fill out the PROMS related to GVHD and sexual function as a screening tool which guide the counselling session and the subsequent genital evaluation. The counselling consists of guidance and follow-up on relevant issues related to disease and treatment sexual complications including genital GVHD. The first intervention visit will be conducted in-person in the outpatient clinic. Subsequent visits can be conducted in-person or over the telephone. Participants with complex sexual health concerns will be referred to the Sexual Health Clinic at Rigshospitalet for further evaluation.

   Genital evaluation Female patients will have a baseline gynecological review with a specialist experienced in post-transplant gynecological care during their preexamination week. During the intervention the patients will have 5 preventive control visits which include a through genital examination and evaluation including menopausal symptoms, genital GVH, and genital tract malignancies.

   Male patients will have a baseline urological review with a specialist experienced in post-transplant urological care. During the intervention the patients will have 5 preventive control visits, and the consultation will include a through genital examination and evaluation including genital GVHD.

   5.6 Data collection

   Participant and disease characteristics will be obtained from the participants. These will include age, gender, marital status, education, employment status, disease type and status, type and intensity of treatment. The patient-reported outcome measure (PROM) include:

   Primary outcome

   • The primary outcome is sexual function which will be assessed by FSFI in female participants, and in male participants by IIEF.

   Secondary outcomes
   * Feasibility of the intervention will be evaluated as acceptability, practicability, integration, adherence to protocol, resource utilization and safety.
   * Sexual distress will be assessed by the FSDS-R.
   * Symptoms of genital GVHD will be assessed by specially developed questions based on clinical and experienced manifestations of genital GVHD.
   * Symptoms of GVHD in other organs will be assessed by the chronic GVHD symptom scale. The scale contains 30 items in 7 subscales (skin, eye, mouth, lung, nutrition, energy, and psychological), and patients report their level of symptom over the past month.
   * Quality of life will be assessed by EORTC-C30.
   * Symptom burden will be assessed with MDASI. 5.7 Analysis Study feasibility parameters will be described and analyzed using descriptive statistics. The demographic and clinical characteristics of participants will be summarized in percentages for categorical variables and mean (SD) for noncategorical variables. Mean score will be calculated for each group and compared using student´s t-test. The domains of questionnaires will be calculated for each group and compared using Wilcoxon´s rank-sum test. Throughout, two-sided P-values <0.05 confidence intervals are considered indicators of statistical significance. Statistical analysis will be conducted using IBM SPSS Statistics for Windows, version 25.

   Sample size
   * In female patients, assuming a difference of size 2.1 for the primary outcome (FSFI) between intervention and control group and a standard deviation of 3.86 points for the primary outcome within each group and with a two-sample t-test with a power of 80 % to detect a significant difference at level 0.05 if 55 patients are included in each treatment arm. To account for an expected dropout rate of 20 % the investigators decided to increase this number to a group size of 66.
   * In male patients, assuming a difference of size 5.0 for the primary outcome (IIEF) between intervention and control group and a standard deviation of 9.3 points for the primary outcome within each group and with a two-sample t-test with a power of 80 % to detect a significant difference at level 0.05 if 56 patients are included in each treatment ar. To account for an expected dropout rate of 20 % the investigators decided to increase this number to a group size of 67.

   There is yearly around 95 patients receiving HSCT at Department of Hematology, Rigshospitalet. Based on this and an expected acceptance of 75%, the investigators aim to include 133 patients in each arm of the study, and therefore the project is estimated to run for 42 months, starting fall 2021.
6. Ethical considerations This study will be registered with the Danish Protection Agency and Clinical Trials. Each participant will receive written and verbal information on the study and assurance of confidentiality according to the principles for research stated in the Helsinki Declaration. Written consent will be obtained from patients participating at time of recruitment. Awareness of the informant's vulnerability mean that additional attention will be paid to the voluntariness in their participation, just as they are given time to debrief and further discuss their experiences.
7. Setting Department of Hematology, Rigshospitalet, Denmark will be Primary sponsor for this project. KHN will be principal investigator of all studies in collaboration with the research management group, the national and international research collaborators (mentors) and clinical collaborators who all have agreed to participate in the study (Figure 2, Table 1).

ELIGIBILITY:
Inclusion Criteria:

* Patients (age>18 years) with a hematologic malignancy who is planned to undergo an HSCT, who provide informed written consent and can understand, speak and read Danish are eligible to participate.

Exclusion Criteria:

* The exclusion criteria include patients with dementia, psychotic disorders, or other cognitive diseases or conditions that hinder participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-11-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
sexual function | 18 month
  The primary outcome is sexual function which will be assessed by Female Sexual Function Index FSFI in female participants
sexual function | 18 month
  The primary outcome is sexual function which will be assessed by The International Index of Erectile Function Questionnaire IIEF in male patients

SECONDARY OUTCOMES:
Evaluation of acceptability of intervention | 18 month
  Feasibility of the intervention will be evaluated as acceptability measured by the rate of included participants, the dropout rate and the rate of completing participants
Evaluation of practicability of intervention | 18 month
  Feasibility of the intervention will be evaluated as practicability measured by logistics or other circumstances challenging adherence during intervention
Evaluation of integration of intervention | 18 month
  Feasibility of the intervention will be evaluated as integration measured by an evaluation of the intergration of the intervention in the clinical praticice and daily work
Evaluation of utilization of intervention | 18 month
  Feasibility of the intervention will be evaluated as resource utilization measured by the total amount of time pr patient of nurse konsultation hours including preparation, and of doctor consultation
Evaluation of safety of intervention | 18 month
  Feasibility of the intervention will be evaluated as safety measured by unexpected adverse events
Evaluation of Sexual distress | 18 month
  Sexual distress will be assessed by the Female Sexual Distress Scale - Revised (FSDS-R) with higher scores indication higher sexual distress.
Description of symptoms of genital GVHD | 18 month
  Symptoms of genital GVHD will be assessed by specially developed questions based on clinical and experienced manifestations of genital GVHD.
Description of symptoms of GHVD | 18 month
  Symptoms of GVHD in other organs will be assessed by the chronic GVHD symptom scale. The scale contains 30 items in 7 subscales (skin, eye, mouth, lung, nutrition, energy, and psychological), and patients report their level of symptom over the past month
Evaluation of quality of life in participants | 18 month
  Quality of life will be assessed by by The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-C30) with higher scores indicating better quality of life.
Evaluation of Symptom burden | 18 month
  Symptom burden will be assessed with M.D. Anderson Symptom Inventory (MDASI) which is a 19 item measure and assesses the severity of 13 symptoms and their impact in cancer patients

CONTACTS AND LOCATIONS:
Locations (1):
- Kristina Nørskov, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Norskov KH, Schjoedt I, Tolver A, Jarden M. Sexual health in patients with malignant hematological disease: a Danish cross-sectional study. Sex Med. 2024 Sep 13;12(4):qfae053. doi: 10.1093/sexmed/qfae053. eCollection 2024 Aug. PMID 39281809